CLINICAL TRIAL: NCT00400738
Title: Pharmacokinetics of and Rate of HIV-1 RNA Decline in ARV-naive HIV-1 Infected Patients Treated With Low- or Standard-dose Saquinavir HGC (Invirase®) and Lopinavir/Ritonavir (Kaletra®
Brief Title: The Pharmacokinetics of Double Boosted Protease Inhibitors in Antiretroviral-naive HIV-1 Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Roche Pharma AG (Industry); International Antiviral Therapy Evaluation Center (Other); Kirby Institute (Other Government)
Responsible Party: Kiat Ruxrungtham, HIV-NAT
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 019
Record Dates: First submitted 2006-11-09; First posted 2006-11-17 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: HIV Infections
Keywords: HIV-1 infection; pharmacokinetics; protease inhibitor; double boosted protease inhibitors; PIs; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Saquinavir; Lopinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): different dose per arm
  Interventions: Drug: Saquinavir, lopinavir, ritonavir
- 2 (Experimental): different dose per arm
  Interventions: Drug: Saquinavir, lopinavir, ritonavir
- 3 (Experimental): different dose per arm
  Interventions: Drug: Saquinavir, lopinavir, ritonavir
- 4 (Experimental): different dose per arm
  Interventions: Drug: Saquinavir, lopinavir, ritonavir

INTERVENTIONS:
Drug: Saquinavir, lopinavir, ritonavir — arm 1 = LPV/RTV 400/100 mg BID + SQV 1000 mg BID arm 2 = LPV/RTV 400/100 mg BID + SQV 600 mg BID arm 3 = LPV/RTV 266/66 mg BID + SQV 1000 mg BID arm 4 = LPV/RTV 266/66 mg BID + SQV 600 mg BID

SUMMARY:
Treatment with only protease inhibitors might benefit HIV patients. Laboratory data have shown that the combination of saquinavir with lopinavir and ritonavir may a good regimen. This study will explore this idea.

DETAILED DESCRIPTION:
Treatment with only protease inhibitors might benefit HIV patients, who experience problems with the other antiretrovirals drugs classes. Another reason to only use protease inhibitors is that the remaining classes are spared. This leaves the option to use these classes in the future, for instance in cases of drug resistance. Laboratory data have shown that the combination of saquinavir with lopinavir and ritonavir may a good regimen. This study will explore this idea.

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent
2. ARV-naïve
3. HIV-1 infected Thai male or female > 18 years old
4. Documented positive test for HIV-1 infection

Exclusion Criteria:

1. Inability to understand the nature and extent of the study and the procedures required.
2. Pregnancy or lactating
3. Active opportunistic infection
4. ALT/ AST more than 2x upper limit
5. creatinine more than 1.5 time the upper limit
6. Smoke cigarettes more than 10 cigarettes a day.
7. Drink alcohol more than 2 units a day
8. Relevant history or current condition, illness that might interfere with drug absorption, distribution, metabolism or excretion.
9. Use of concomitant medication that may interfere with the pharmacokinetics of lopinavir/ritonavir or saquinavir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
study the pharmacokinetics of low dose and standard dose lopinavir/ritonavir and saquinavir HGC in ARV naive HIV-1 infected Thai patients | 1 year

SECONDARY OUTCOMES:
To describe short-term tolerability, toxicity and efficacy of combinations of low-dose and standard dose lopinavir/ritonavir and saquinavirHGC given to the patients in this trial | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrunghtam, MD, PhD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration; Joep Lange, MD, PhD, Study Chair — International Antiviral Therapy Evaluation Center (IATEC), Center for Poverty-related Communicable Diseases, Department of Internal Medicine, Academic Medical Center (AMC), University of Amsterdam (UVA); Praphan Phanuphak, MD, PhD, Study Chair — The HIV Netherlands Australia Thailand Research Collaboration; David Burger, PharmD, PhD, Study Chair — Radboud University Medical Center; David Cooper, MD, PhD, Study Chair — National Center in HIV Epidemiology and Clinical Research
Locations (1):
- The HIV Netherlands Australia Thailand Research Collaboration, Bangkok, Thailand

REFERENCES:
- [Background] van der Lugt J, Autar RS, Ubolyam S, Garcia EF, Sankote J, Avihingsanon A, Chuenyam T, Cooper DA, Lange J, Phanuphak P, Wit F, Ruxrungtham K, Burger D; HIV-NAT 019 Study Team. Pharmacokinetics and short-term efficacy of a double-boosted protease inhibitor regimen in treatment-naive HIV-1-infected adults. J Antimicrob Chemother. 2008 May;61(5):1145-53. doi: 10.1093/jac/dkn050. Epub 2008 Feb 18. PMID 18285316
- [Derived] Maughan RT, Feeney ER, Capel E, Capeau J, Domingo P, Giralt M, Lange JM, Phanuphak P, Cooper DA, Reiss P, Mallon PW; HIVNAT-019 Study Group. Improved adipose tissue function with initiation of protease inhibitor-only ART. J Antimicrob Chemother. 2016 Nov;71(11):3212-3221. doi: 10.1093/jac/dkw301. Epub 2016 Aug 11. PMID 27516476